CLINICAL TRIAL: NCT06162910
Title: Aspiration Risk in Stroke Units. Validation of Clinical Investigation Procedures for Risk Stratification
Brief Title: Validation of Aspiration Risk Assessment in Stroke Units
Acronym: ARAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis resulted in reliable figures
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ARAS-1
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical swallowing exam (Experimental): Patients with acute ischemic stroke
  Interventions: Diagnostic Test: Daniels Water Swallow Test; Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Diagnostic Test: Daniels Water Swallow Test — Clinical water swallow dysphagia screening
Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing — Endoscopic evaluation of swallowing function
  Other Names: FEES

SUMMARY:
The purpose of the study is to test the validity of a modified Daniels swallow test. The original test serves as reference method, the swallow endoscopy (FEES) as "gold standard".

Furthermore, it will be examined whether the modified Daniels test can be performed by nursing staff. As a reference method, the test will be performed by experienced speech therapists and the swallowing endoscopy (FEES) by speech therapists and/or physicians.

DETAILED DESCRIPTION:
For each included patient, the standardized Daniels test is performed by a speech therapist within the first 24 hours after admission, as well as the modified Daniels test by a second speech therapist who is blinded to the result of the first test. This is immediately followed by the administration of the modified Daniels test by a nurse. All investigators are blinded to the results of the preceding water swallow tests. The water swallow tests are not performed by physicians.

Following the water swallow tests, FEES is performed by an examiner (physician or speech therapist) experienced in FEES. The examination is digitally recorded and evaluated by an external examiner (physician or speech therapist) using validated scores.

ELIGIBILITY:
Inclusion Criteria:

* Acute (maximum 7 days old) cerebral infarction detected by cMRI or cCT
* Neurological deficits
* Written informed consent

Exclusion Criteria:

* Cerebral hemorrhage
* Pre-existing swallowing disorders of other etiologies
* Contraindications to clinical swallowing examination (lack of alertness as well as lack of compliance) - Contradictions to FEES (lack of alertness as well as lack of compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration-Score (PAS) Penetration-Aspiration-Score (PAS) | Immediately after the intervention
  Penetration-Aspiration-Score, minimum value 1, maximum value 8; higher scores mean worse outcome

SECONDARY OUTCOMES:
Functional Oral Intake Scale-German (FOIS-G) | Immediately after the intervention
  Functional Oral Intake Scale - German Version; minimum value 1, maximum value 7; higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Samra Hamzic, PhD, Principal Investigator — University Hospital Giessen and Marburg, Campus Giessen; Tobias Braun, MD, Study Director — University Hospital Giessen and Marburg, Campus Giessen
Locations (1):
- University Hospital Giessen and Marburg, Campus Giessen, Giesen, Hesse, Germany